CLINICAL TRIAL: NCT06556381
Title: The Efficacy of Ultrasound-guided Transversus Abdominis Plane ( TAP) Block Versus Standard Analgesic Protocol for Postoperative Analgesia After Elective, Cesarean- Section Delivery- A Randomize Controlled Trial
Brief Title: Efficacy of Trans Abdominis Plane Block for Post Cesarean Delivery Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Mohammed Abaalkhayl, Associate Proffesor, Qassim University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 607/46/828
Record Dates: First submitted 2024-08-01; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Analgesia
Keywords: Pain; cesarean delivery
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A, (Experimental): women who received TAP block.
  Interventions: Procedure: TAP block
- Group B (Active Comparator): Received Usual modality of analgesics (Paracetamol, Tramadol, and Pethidine).
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: TAP block — Women will receive TAP block.

SUMMARY:
Relief from pain is part of the fundamental human right to health. (1) However, available evidence indicates an increasingly detailed understanding of the pathophysiology of pain and general inadequacy of its treatment.

DETAILED DESCRIPTION:
Background: Relief from pain is part of the fundamental human right to health. (1) However, available evidence indicates an increasingly detailed understanding of the pathophysiology of pain and general inadequacy of its treatment.

Rationale: Assessment and Improving the Pain Management Modality

Study objectives: In this study, determined the efficacy of TAP block in patients undergoing cesarean section.

Methods:

This study is a cross-sectional study. It is a multi-centric study as it was conducted in different Governmental hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-50 years
2. Patients of >50 kg or <100 kg weight.
3. Urgency: Elective, Emergent and Urgent cases

Exclusion Criteria:

1. Patients of <50 kg or >100 kg weight
2. Any contraindication to any of anesthesia medications
3. Patient unable to understand numeric rating scale (NRS)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 24 hours
  NRS

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abaalkhayl, MD, Principal Investigator — Qassim University
Locations (1):
- Qassim University Medical City, Buraidah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided